CLINICAL TRIAL: NCT00034684
Title: Safety and Tolerability Study of Farnesyl Protein Transferase Inhibitor (FPTI) in Patients With Leukemia
Brief Title: Study of Farnesyl Protein Transferase Inhibitor (FPTI) in Patients With Leukemia (Study P00701)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00701
Record Dates: First submitted 2002-05-01; First posted 2002-05-02 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic; Blast Crisis; Leukemia, Lymphocytic
Keywords: Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid; Leukemia, Lymphocytic
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis; Leukemia, Lymphoid; Leukemia, Myeloid | interventions — 2-(2-oxo-2-((3,7,11-trimethyl-2,6,10-dodecatrienyl)oxy)aminoethyl)phosphonic acid, (2,2-dimethyl-1-oxopropoxy)methyl ester sodium

INTERVENTIONS:
Drug: Farnesyl Protein Transferase Inhibitor

SUMMARY:
The purpose of this study is to determine the safety and tolerability of an oral Farnesyl Protein Transferase Inhibitor (SCH 66336) as a single agent in patients with Advanced Myelodysplastic Syndrome, Acute Myelogenous Leukemia, Chronic Myelogenous Leukemia in Blast Crisis, or Acute Lymphoblastic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically documented chronic myelogenous leukemia in blast crisis, myelodysplasia, acute myelogenous leukemia, or acute lymphocytic leukemia.
* Life expectancy of 12 weeks or greater.
* ECOG Performance Status less than or equal to 2.
* Meets protocol requirements for specified laboratory values.
* No manifestations of a malabsorption syndrome.

Exclusion Criteria:

* Patients who have received more than three chemotherapy regimens for more than three recurrences of the disease.
* Poor medical risks because of nonmalignant systemic disease as well as those with active uncontrolled conditions.
* Patients who have received investigational therapy of any type within 30 days prior to administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2001-07; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)